CLINICAL TRIAL: NCT04582591
Title: A Phase II Trial of Cannabidiol for Prevention of Chemotherapy-induced Peripheral Neuropathy in Patients Receiving Oxaliplatin or Paclitaxel Based Chemotherapy
Brief Title: Cannabidiol for Prevention of Chemotherapy-induced Peripheral Neuropathy
Acronym: CINCAN-2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zealand University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REG-114-2020
Record Dates: First submitted 2020-09-29; First posted 2020-10-09 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2021-07

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: CIPN; Cannabinoid; Cannabidiol; CBD; Neurotoxic Chemotherapy; paclitaxel; oxaliplatin; Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cannabidiol (Experimental): Patients will receive cannabidiol in conjunction with their standard chemotherapy treatment
  Interventions: Drug: Cannabidiol 100 MG/ML

INTERVENTIONS:
Drug: Cannabidiol 100 MG/ML — Patients receive cannabidiol before and after treatment with chemotherapy
  Other Names: CBD

SUMMARY:
This protocol describes a phase II trial investigating the efficacy of CBD in paclitaxel- and oxaliplatin-induced peripheral neuropathy. The trial uses multiple assessments such as validated PRO-questionnaires and multifrequency vibrometry.

DETAILED DESCRIPTION:
Chemotherapy induced peripheral neuropathy (CIPN) is among the most feared side effects to cancer treatment. The development of CIPN can lead to omission or even discontinuation of antineoplastic drugs, possibly affecting efficacy of cancer treatment. There is a lack of knowledge about the natural course of CIPN and to this date, there are no available methods for the early detection of CIPN. With no effective prevention or treatment options, the condition has severe impact on patient quality of life and healthcare expenditure.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* A diagnosis of cancer.
* Fulfill criteria for starting chemotherapy.
* Scheduled to undergo at least 6 courses of paclitaxel or 4 courses of oxaliplatin based chemotherapy.
* If not postmenopausal (defined as no menses for 12 months without an alternative medical cause), women will have use effective anti-contraception (using definitions in the CTFG*-Recommendations related to contraception and pregnancy testing in clinical trials) and submit to a monthly pregnancy test (blood test).

Exclusion Criteria:

* Unable to complete PRO-measurements.
* Previously received taxanes or platinum-based chemotherapy.
* If using any antiepileptic or antidepressant medicine (ATC: N03A or N06A). Treatment must be stable (no changes in dosing in last 30 days) prior to inclusion. However, any treatment with Clobazam (N05BA09) is not allowed due to major interaction with cannabidiol.
* Use of cannabinoids. If in use, treatment must be stopped 4 days prior to inclusion.
* Hypersensitivity reactions towards Ascorbylpalmitat or Triglycerides (medium-chain)
* Baseline transaminase level must not be above 3 times the Upper Limit of Normal (ULN) at study beginning.
* Women who are breastfeeding.
* Concomitant treatment with strong inducers of CYP3A4 and/or strong inducers of CYP2C19.

CTFG: The Heads of Medicines Agencies commissioned Clinical Trials Facilitation Group under the European Union's clinical trials directive 2001/20.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Difference in Acute Neuropathic Symptoms from baseline and during 1. course chemotherapy. | up to 5 days
  Difference in the North Central Cancer Treatment Group (NCCTG)- acute-CIPN Questionnaire from baseline compared to 3-5 days after initiation of chemotherapy course no. 1.
  The Questionnaire contains single items questions, answerable on a 0-10 numeric scale, 0 corresponds to no symptoms and 10 worst possible symptoms.
Difference in Vibrograms from baseline and during 1. course chemotherapy. | up to 5 days
  Difference in the Vibrograms from baseline compared to 3-5 days after initiation of chemotherapy course no. 1.

SECONDARY OUTCOMES:
Difference in baseline vibrograms of patients treated with CBD compared to vibrograms at follow-up 3 mo. after the end of the 6th course of chemotherapy or the last course of chemotherapy (if before course no. 6). | through study completion, an average of 1 year and 6 months
  For patients receiving paclitaxel-based chemotherapy
Difference in baseline vibrograms of patients treated with CBD compared to vibrograms at follow-up 3 mo. after the end of the 4th course of chemotherapy or the last course of chemotherapy (if before course no. 4) | through study completion, an average of 1 year and 6 months
  For patients receiving oxaliplatin-based chemotherapy
Difference in CIPN from baseline to after chemotherapy course no. 3 | through study completion, an average of 1 year and 6 months
  For patients receiving paclitaxel: Difference in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Chemotherapy-induced Peripheral Neuropathy Questionnaire Module (EORTC-QLQ-CIPN20) from baseline compared to after chemotherapy course no. 3.
  The EORTC-QLQ-CIPN20 is a validated 20-item patient reported outcome questionnaire. Items are answered on a scale from 1-4. 1 corresponds to no symptoms and 4 to "a lot" of symptoms. A summary score will be calculated based on items 1-18, Min. value 18, Max. value 72.
Difference in CIPN from baseline to after chemotherapy course no. 6 | through study completion, an average of 1 year and 6 months
  For patients receiving paclitaxel: Difference in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Chemotherapy-induced Peripheral Neuropathy Questionnaire Module (EORTC-QLQ-CIPN20) EORTC-QLQ-CIPN20 from baseline compared to after chemotherapy course no. 6.
  The EORTC-QLQ-CIPN20 is a validated 20-item patient reported outcome questionnaire. Items are answered on a scale from 1-4. 1 corresponds to no symptoms and 4 to "a lot" of symptoms. A summary score will be calculated based on items 1-18, Min. value 18, Max. value 72.
Difference in CIPN from baseline to 1. follow-up (PAC) | through study completion, an average of 1 year and 9 months
  For patients receiving paclitaxel: Difference in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Chemotherapy-induced Peripheral Neuropathy Questionnaire Module (EORTC-QLQ-CIPN20) from baseline compared to 1. Follow-up, 3 mo. after chemotherapy.
  The EORTC-QLQ-CIPN20 is a validated 20-item patient reported outcome questionnaire. Items are answered on a scale from 1-4. 1 corresponds to no symptoms and 4 to "a lot" of symptoms. A summary score will be calculated based on items 1-18, Min. value 18, Max. value 72.
Difference in CIPN from baseline to after chemotherapy course no. 2 | through study completion, an average of 1 year and 6 months
  For patients receiving oxaliplatin: Difference in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Chemotherapy-induced Peripheral Neuropathy Questionnaire Module (EORTC-QLQ-CIPN20) from baseline compared to after chemotherapy course no. 2.
  The EORTC-QLQ-CIPN20 is a validated 20-item patient reported outcome questionnaire. Items are answered on a scale from 1-4. 1 corresponds to no symptoms and 4 to "a lot" of symptoms. A summary score will be calculated based on items 1-18, Min. value 18, Max. value 72.
Difference in CIPN from baseline to after chemotherapy course no. 4 | through study completion, an average of 1 year and 6 months
  For patients receiving oxaliplatin: Difference in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Chemotherapy-induced Peripheral Neuropathy Questionnaire Module (EORTC-QLQ-CIPN20) from baseline compared to after chemotherapy course no. 4.
  The EORTC-QLQ-CIPN20 is a validated 20-item patient reported outcome questionnaire. Items are answered on a scale from 1-4. 1 corresponds to no symptoms and 4 to "a lot" of symptoms. A summary score will be calculated based on items 1-18, Min. value 18, Max. value 72.
Difference in CIPN from baseline to 1. follow-up (OX) | through study completion, an average of 1 year and 9 months
  For patients receiving oxaliplatin: Difference in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Chemotherapy-induced Peripheral Neuropathy Questionnaire Module (EORTC-QLQ-CIPN20) from baseline compared to 1. Follow-up, 3 mo. after chemotherapy.
  The EORTC-QLQ-CIPN20 is a validated 20-item patient reported outcome questionnaire. Items are answered on a scale from 1-4. 1 corresponds to no symptoms and 4 to "a lot" of symptoms. A summary score will be calculated based on items 1-18, Min. value 18, Max. value 72.
Difference in QoL from baseline to after chemotherapy course no. 3 | through study completion, an average of 1 year and 6 months
  For patients receiving paclitaxel: Difference in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30) from baseline compared to after chemotherapy course no. 3.
  The EORTC-QLQ-C30 is a fully validated and internationally accredited 30-item questionnaire measuring 16 subscales. Items are answered on a scale from 1-4, 1 corresponds to no symptoms and 4 to "a lot" of symptoms. We calculate and report on all 16 subscales.
Difference in QoL from baseline to after chemotherapy course no. 6. | through study completion, an average of 1 year and 6 months
  For patients receiving paclitaxel: Difference in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30) from baseline compared to after chemotherapy course no. 6.
  The EORTC-QLQ-C30 is a fully validated and internationally accredited 30-item questionnaire measuring 16 subscales. Items are answered on a scale from 1-4, 1 corresponds to no symptoms and 4 to "a lot" of symptoms. We calculate and report on all 16 subscales.
Difference in QoL from baseline to after chemotherapy course no. 2 | through study completion, an average of 1 year and 6 months
  For patients receiving oxaliplatin: Difference in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30) from baseline compared to after chemotherapy course no. 2.
  The EORTC-QLQ-C30 is a fully validated and internationally accredited 30-item questionnaire measuring 16 subscales. Items are answered on a scale from 1-4, 1 corresponds to no symptoms and 4 to "a lot" of symptoms. We calculate and report on all 16 subscales.
Difference in QoL from baseline to after chemotherapy course no. 4 | through study completion, an average of 1 year and 6 months
  For patients receiving oxaliplatin: Difference in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30) from baseline compared to after chemotherapy course no. 4.
  The EORTC-QLQ-C30 is a fully validated and internationally accredited 30-item questionnaire measuring 16 subscales. Items are answered on a scale from 1-4, 1 corresponds to no symptoms and 4 to "a lot" of symptoms. We calculate and report on all 16 subscales.
Difference in the Vibrograms after chemotherapy course 1 | through study completion, an average of 1 year and 6 months
  For patients receiving paclitaxel: Difference in the Vibrograms from baseline compared to after chemotherapy course no. 6.
Difference in the Vibrograms after chemotherapy course 2 | through study completion, an average of 1 year and 6 months
  For patients receiving oxaliplatin: Difference in the Vibrograms from baseline compared to after chemotherapy course no. 4.
Dose reductions | through study completion, an average of 1 year and 6 months
  Number of patients needing a dose reduction in accordance with national Danish treatment guidelines(reasons for discontinuation will be registered).
Dose delays | through study completion, an average of 1 year and 6 months
  Number of patients needing a dose delay in accordance with national Danish treatment guidelines(reasons for discontinuation will be registered).
Not completing planned courses of chemotherapy | through study completion, an average of 1 year and 6 months
  Number of patients not completing their planned courses of chemotherapy (reasons for discontinuation will be registered).

OTHER OUTCOMES:
Side Effects (Clinician Scored) | through study completion, an average of 1 year and 6 months
  Side effects will be registered and scored according to the Common Terminology Criteria for Adverse Events v4.03 (CTCAE v4.03).
  The CTCAE grades side effects on a 1-5 scale. 1 represents best symptom manifestation and 5 represents death from specific side effect.
Side Effects (Patient Reported) | through study completion, an average of 1 year and 6 months
  Patients will be asked to report their side effects using an digitalized version of the Patient Reported Outcome of Common Terminology Criteria for Adverse Events. (PRO-CTCAE).
  The PRO-CTCAE items evaluate different symptom attributes; frequency, severity, interference, amount, presence/absence, utilizing "yes" and "no" categories for presence/absence and a 1-5 grading scale for frequency, severity, interference, amount. 1 corresponds to best symptoms manifestation, 5 to worst symptom manifestation.
Change in vibrograms at day 3-5 from baseline compared to overall CIPN18 score at 3 months (PAC) | through study completion, an average of 9 months
  For patients receiving paclitaxel: Difference in the Vibrograms at day 3-5 from baseline compared to CIPN18 total score at follow-up 3 months after treatment
Change in vibrograms at day 3-5 from baseline compared to overall CIPN18 score at 3 months (OX) | through study completion, an average of 9 months
  For patients receiving oxaliplatin: Difference in the Vibrograms at day 3-5 from baseline compared to CIPN18 total score at follow-up 3 months after treatment
Change in vibrograms at day 3-5 from baseline compared to overall CIPN18 score at 12 months (PAC) | through study completion, an average of 1 year and 6 months
  For patients receiving paclitaxel: Difference in the Vibrograms at day 3-5 from baseline compared to CIPN18 total score at follow-up 12 months after treatment
Change in vibrograms at day 3-5 from baseline compared to overall CIPN18 score at 12 months (OX) | through study completion, an average of 1 year and 6 months
  For patients receiving oxaliplatin: Difference in the Vibrograms at day 3-5 from baseline compared to CIPN18 total score at follow-up 12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jørn Herrstedt, DMSc, Study Chair — Zealand University Hospital / University of Copenhagen; Sebastian W Nielsen, MD, Principal Investigator — Zealand University Hospital / University of Copenhagen
Locations (1):
- Department of Clinical Oncology and Palliative Care, Roskilde, Denmark

IPD SHARING:
Plan to Share IPD: No